CLINICAL TRIAL: NCT07366112
Title: CDK4/6 Inhibitors Combined With Endocrine Therapy for Neoadjuvant Treatment of Breast Cancer: ctDNA-Guided Personalized Therapy
Brief Title: CDK4/6 Inhibitors Combined With Endocrine Therapy for Neoadjuvant Treatment
Acronym: DNACDKHR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Shu Wang, director of breast center, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH2025CDK46NAE
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hormone Receptor-Positive Breast Cancer; High-risk Breast Cancer; Early-Stage Breast Cancer; HER2-negative Breast Cancer; ctDNA Monitoring
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients receives oral CDK4/6 inhibitor combined with endocrine therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CDK4/6 inhibitor with endocrine therapy (Experimental): Patients receive 4 cycles of neoadjuvant CDK4/6 inhibitor with endocrine therapy. Post-surgery treatment is guided by ctDNA status:
  ctDNA-negative at baseline and post-neoadjuvant, with post-op Ki67 ≤10% ：Continue CDK4/6 inhibitor with endocrine therapy for 2-3 years.
  ctDNA-positive → negative, or persistently ctDNA-negative with post-op Ki67 >10% :
  Randomized 1:1 to:
  Arm 1: CDK4/6 inhibitor with endocrine therapy for 2-3 years. Arm 2: Adjuvant chemotherapy (investigator's choice) → CDK4/6 inhibitor with endocrine therapy for 2-3 years.
  （3）Persistently ctDNA-positive or ctDNA-negative → positive: Adjuvant chemotherapy → CDK4/6 inhibitor with endocrine therapy for 2-3 years.
  Premenopausal women receive ovarian suppression with LHRH agonists.
  Interventions: Drug: CDK4/6 inhibitor with endocrine therapy

INTERVENTIONS:
Drug: CDK4/6 inhibitor with endocrine therapy — CDK4/6 inhibitor with endocrine therapy for neoadjuvent therapy

SUMMARY:
Exploring the dynamics of ctDNA following neoadjuvant therapy with CDK4/6 inhibitors combined with endocrine treatment, and its potential to guide de-escalation of adjuvant chemotherapy

DETAILED DESCRIPTION:
Breast cancer remains a leading cause of cancer-related morbidity and mortality globally, with hormone receptor-positive (HR+), HER2-negative (HER2-) subtypes accounting for approximately 70% of cases. While adjuvant chemotherapy is standard for high-risk early-stage HR+/HER2- breast cancer, it carries significant toxicity, and many patients may not derive clinical benefit. Emerging evidence suggests that circulating tumor DNA (ctDNA)-a minimally invasive biomarker reflecting residual disease-may guide personalized treatment de-escalation.

Preclinical and clinical studies demonstrate that ctDNA dynamics correlate with tumor burden and prognosis. In HR+ breast cancer, ctDNA clearance after neoadjuvant therapy is associated with improved survival, while persistent ctDNA post-treatment predicts recurrence. CDK4/6 inhibitors, such as Dalpiciclib, have revolutionized advanced HR+/HER2- breast cancer management by enhancing endocrine therapy efficacy. However, their role in early-stage disease, particularly in a ctDNA-guided de-escalation strategy, remains underexplored. This study addresses this gap by evaluating whether ctDNA-driven decision-making can safely reduce chemotherapy use while maintaining clinical outcomes.

Study Objectives Primary Objectives: Assess ctDNA clearance rate (defined as conversion from detectable to undetectable ctDNA) after 4 cycles of neoadjuvant CDK4/6i + endocrine therapy.

Secondary Objectives Evaluate 3-year event-free survival (EFS), where events include local/distant recurrence, secondary malignancies, or death.

Compare safety profiles of CDK4/6i + endocrine therapy versus chemotherapy.

Evaluate tumor response metrics:

Pathological complete response (pCR) and residual cancer burden (RCB 0-1). Complete cell cycle arrest (CCCA; Ki67 ≤2.7%). Assess objective response rate (ORR) by RECIST 1.1.

Exploratory Objectives Correlate ctDNA clearance with long-term outcomes (e.g., EFS, overall survival).

Study Design

All patients received 4 cycles of neoadjuvant CDK4/6i + endocrine therapy. Post-Surgery Treatment： ctDNA-negative post-neoadjuvant: Continue CDK4/6i + endocrine therapy ctDNA-positive post-neoadjuvant: Optional adjuvant chemotherapy followed by CDK4/6i + endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1.Female breast cancer patients aged ≥18 years and ≤75 years, either postmenopausal or premenopausal/perimenopausal; 2.Pathologically confirmed hormone receptor-positive (HR+), HER2-negative invasive breast cancer:

  1. ER-positive and/or PR-positive defined as: ≥10% of tumor cells showing positive staining;
  2. HER2-negative defined as: standard immunohistochemistry (IHC) result of 0/1+; or IHC 2+ with negative in situ hybridization (ISH) (confirmed by the central pathology laboratory); 3. At least one evaluable lesion per RECIST 1.1, with clinical staging meeting:

  <!-- -->

  1. T1c-2N0M0 with high-risk factors (Grade 3, or Grade 2 with Ki67 ≥20%);
  2. T3N0M0;
  3. Any TN+M0; 4.Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1; 5.Willing to participate in the study and voluntarily sign informed consent; 6.Agree to undergo ctDNA testing during treatment; 7.Adequate organ and bone marrow function defined as:

  <!-- -->

  1. Absolute neutrophil count (ANC) ≥1,500/mm³ (1.5 × 10⁹/L) (without granulocyte colony-stimulating factor [G-CSF] treatment within 14 days);
  2. Platelet count (PLT) ≥100,000/mm³ (100 × 10⁹/L) (without corrective therapy within 7 days);
  3. Hemoglobin (Hb) ≥9 g/dL (90 g/L) (without corrective therapy within 7 days);
  4. Serum creatinine ≤1.5× upper limit of normal (ULN) or creatinine clearance ≥60 mL/min (without corrective therapy within 7 days);
  5. Total bilirubin (TBIL) ≤1.5×ULN (without corrective therapy within 7 days);
  6. Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤1.5×ULN (without corrective therapy within 7 days);
  7. Cardiac function: left ventricular ejection fraction (LVEF) ≥55%; QTc interval corrected by Fridericia's formula (QTcF) <470 msec on 12-lead ECG; Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to randomization and agree to use non-hormonal contraception from informed consent signing until 2 months after the last treatment.

Exclusion Criteria:

* 1.Bilateral breast cancer; 2.Prior history of breast cancer (including ductal carcinoma in situ or invasive breast cancer); 3.Any prior antitumor therapy for the current breast cancer, including systemic therapies (endocrine, chemotherapy, immunotherapy, biological therapy) or local therapies (radiotherapy, vascular embolization, axillary lymph node biopsy); 4.Diagnosis of any malignancy within 5 years prior to randomization, except cured cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma of the skin; 5.History of severe pulmonary diseases (e.g., interstitial pneumonia); 6. HIV infection, acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA ≥500 IU/mL), hepatitis C (HCV antibody-positive with HCV RNA above the lower limit of detection), or co-infection with HBV and HCV; 7.Within 6 months prior to randomization: myocardial infarction, severe/unstable angina, NYHA Class ≥II heart failure, ≥Grade 2 persistent arrhythmia (per NCI CTCAE v5.0), atrial fibrillation of any grade, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident (including transient ischemic attack), or symptomatic pulmonary embolism; 8.Severe active infection within 4 weeks prior to randomization (requiring intravenous antibiotics, antifungals, or antivirals) or unexplained fever >38.5°C during screening/before first dose; 9.Known allergy to any component of the study drugs; 10.Current participation in another interventional drug clinical study; 11.Pregnancy or lactation; 12.Refusal to comply with follow-up; 13.Other severe physical/mental illnesses or laboratory abnormalities that may increase study risk, interfere with results, or render the patient unsuitable per investigator judgment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
ctDNA Clearance Rate after Neoadjuvant Therapy | From baseline to 4 weeks post-neoadjuvant therapy (pre-surgery)
  Proportion of patients achieving conversion from detectable to undetectable ctDNA in plasma after 4 cycles of neoadjuvant CDK4/6i+endocronetherapy. ctDNA analysis uses tumor-informed personalized panels (tracking 16 clonal variants via whole-exome sequencing), with clearance defined as ≥2 consecutive negative results at 1% variant allele frequency threshold.

SECONDARY OUTCOMES:
3-Year Event-Free Survival (EFS) | From neoadjuvant therapy to 36 months post-surgery
  Time from randomization to first occurrence of locoregional/distant recurrence, contralateral breast cancer, secondary malignancy, or death from any cause. Assessed via imaging (CT/MRI), pathology, and clinical exams every 3 months for 3 years. Events are adjudicated by blinded independent review committee.
Residual Cancer Burden (RCB) 0-1 Rate | At surgery (approximately 16 weeks since neoadjuvant therapy)
  Proportion of patients achieving RCB 0 (pathological complete response) or RCB-1 (minimal residual disease) in surgical specimens. RCB is calculated using standardized criteria (tumor bed area, cellularity, nodal involvement) by blinded central pathology review.
Objective Response Rate (ORR) by RECIST 1.1 | Baseline to pre-surgery (week 16)
  Proportion of patients with complete/partial response per RECIST 1.1 criteria during neoadjuvant phase, measured by MRI/CT. Target lesion size reduction ≥30% (partial) or disappearance (complete) required, confirmed by two consecutive assessments ≥4 weeks apart.
Complete Cell Cycle Arrest (CCCA) Rate (Ki67 ≤2.7%) | Post-neoadjuvant therapy (pre-surgery, week 16)
  Percentage of patients with Ki67 ≤2.7% in post-neoadjuvant tumor biopsies, assessed via immunohistochemistry (IHC) with 3,3'-diaminobenzidine staining. Central laboratory quantification uses Aperio image analysis system (Leica Biosystems).
Incidence of Grade ≥3 Treatment-Related Adverse Events (TRAEs) | From first dose to 30 days after last treatment
  Proportion of patients experiencing grade ≥3 adverse events (per NCI CTCAE v5.0) related to Dalpiciclib + AI or chemotherapy, including hematologic (neutropenia, anemia), hepatic (ALT/AST elevation), and cardiac (LVEF decline ≥10%) toxicities. Events are monitored every cycle during neoadjuvant therapy and quarterly during adjuvant phase.

CONTACTS AND LOCATIONS:
Overall Officials: shu wang, doctor, Principal Investigator — Peking University People's Hospital